CLINICAL TRIAL: NCT05666869
Title: Tolerance Assesment of the Usage of an Analgesic Dose of Esketamine for Treatment of Moderate to Intense Pain in an Emergency Departement
Acronym: ESKETAMINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association pour la Formation l'Enseignement et la Recherche du Service de l'Accueil des Urgences (Other)
Responsible Party: Sponsor
Other Study IDs: AFERSAU-2022-01
Record Dates: First submitted 2022-12-13; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Pain, Acute
Keywords: analgesia; emergency department; esketamine
MeSH Terms: conditions — Acute Pain; Agnosia; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Esketamine perfusion — Analgesic dose of ESKETAMINE via a 30 minutes.intravenous perfusion

SUMMARY:
KETAMINE has been used for several years in emergency departments for analgesic purposes. Its ease of use and its analgesic effect have been demonstrated in several studies.

Nevertheless, this molecule is not devoid of side effects, in particular the very frequent occurrence of nausea, vomiting, anxiety, an overall feeling of discomfort and more rarely hallucinations, feelings of unreality, or tachycardia.

Recently, ESKETAMINE, used as an anesthetic but also in the USA as an antidepressant, has obtained its Marketing Authorization in the management of moderate to severe pain. ESKETAMINE corresponds to the S-(-)-KETAMINE enantiomer. Like KETAMINE, it acts as a non-competitive antagonist of the N-methyl-D-aspartate (NMDA) receptor but unlike KETAMINE does not interact, with the sigma receptors responsible for hallucinations and delusional symptoms. ESKETAMINE aimed at anesthetic is about twice as potent as KETAMINE and would also be eliminated more quickly.

Studies suggest that at equivalent doses, ESKETAMINE would be better tolerated than the KETAMINE usually used in emergency departments.

In this study, the tolerance of ESKETAMINE used at analgesic doses for treatment of moderate to severe pain will be assessed in an emergency departement

A wider usage of ESKETAMINE for analgesia purpose in emergency departments is expected, with a better tolerance for the patients compared to KETAMINE

ELIGIBILITY:
Inclusion Criteria:

* Age is 18 years old or more
* Moderate to severe pain as assessed by the patient with a verbal numerical rating scale (NRS) of 6/10 or more ; NRS goes from 0 (no pain) to 10 (the worst pain imaginable)
* Physician has decided to use ESKETAMINE
* Patient is not opposed to enroll in the study after having been informed, as attested by the physician in the patient's file

Exclusion Criteria:

* Adult under juridic protection, under guardianship, under curatorship
* Patient unable to express his consent
* Patient deprived of liberty by a judicial or administrative decision
* Pregnant, parturient or nursing mother
* Patients physically or mentally unable to answer the questionnaire
* Typical kidney colic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the emergency department of the university hospital of Nice, France (Hôpital Pasteur 2) from monday to friday, 8h30 am to 6h30 pm, meeting the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
ESKETAMINE adverse reactions | From beginning of perfusion (T0) to patient exit of the emergency department (up to 4 hours after T0)
  Enumeration of the adverse reactions occuring to the patient as collected by the investigator in the patient file and by the patient in the study questionnaire

SECONDARY OUTCOMES:
Pain self assesment T0(a) | beginning of perfusion (T0)
  Numerical pain rating scale spanning from 0 (no pain) to 10 (the worst pain imaginable)
Pain self assesment T0(b) | beginning of perfusion (T0)
  4 points Likert pain relief scale : completely relieved ; much relieved ; a little relieved ; not relieved at all
Pain self assesment T15(a) | 15 minutes after the beginning of perfusion (T0 + 15 minutes)
  Numerical pain rating scale spanning from 0 (no pain) to 10 (the worst pain imaginable)
Pain self assesment T15(b) | 15 minutes after the beginning of perfusion (T0 + 15 minutes)
  4 points Likert pain relief scale : completely relieved ; much relieved ; a little relieved ; not relieved at all
Pain self assesment T30(a) | 30 minutes after the beginning of perfusion (T0 + 30 minutes)
  Numerical pain rating scale spanning from 0 (no pain) to 10 (the worst pain imaginable)
Pain self assesment T30(b) | 30 minutes after the beginning of perfusion (T0 + 30 minutes)
  4 points Likert pain relief scale : completely relieved ; much relieved ; a little relieved ; not relieved at all
Patient satisfaction about his treatment (T15) | 15 minutes after the beginning of perfusion (T0 + 15 minutes)
  Self assessed 3 points Likert satisfaction scale : Very satisfied; Satisfied ; Not satisfied
Patient satisfaction about his treatment (T30) | 30 minutes after the beginning of perfusion (T0 + 30 minutes)
  Self assessed 3 points Likert satisfaction scale : Very satisfied; Satisfied ; Not satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Julie Contenti, MD, PhD, Study Director — Association pour la Formation l'Enseignement et la Recherche du Service de l'Accueil des Urgences
Locations (1):
- Centre Hospitalier Universitaire de Nice, Nice, Alpes Maritimes, France